CLINICAL TRIAL: NCT05468840
Title: A Double Blinded, Randomized, Placebo Controlled, Parallel Arm Pilot Trial of Intravenous Ketamine for Emergency Department Treatment of Suicidal Ideation in a Pediatric Population
Brief Title: Study of IV Ketamine for Emergency Department Treatment of Adolescent Suicidal Ideation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Michael Schlegelmilch, Principal Investigator, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0000001
Record Dates: First submitted 2022-07-11; First posted 2022-07-21 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Suicidal Ideation
Keywords: ketamine; emergency department; pediatrics
MeSH Terms: conditions — Suicidal Ideation; Emergencies | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intravenous ketamine infusion (Experimental): Participants in the intervention group will receive 0.5mg/kg of 1mg/mL intravenous ketamine (50 mg maximum) over 40 minutes.
  Interventions: Drug: Ketamine Hydrochloride
- Intravenous normal saline infusion (Placebo Comparator): Participants in the control group will receive 0.5mL/kg intravenous normal saline (50 ml maximum) over 40 minutes.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ketamine Hydrochloride — see study arm description
  Other Names: ketamine
  Arms: Intravenous ketamine infusion
Drug: Normal saline — see study arm description
  Arms: Intravenous normal saline infusion

SUMMARY:
Approximately 20% of Canadian adolescents experience thoughts of suicide, or suicidal ideation (SI), and suicide is the second leading cause of death among Canadians aged 15-19 years. The emergency department at CHEO sees approximately four patients per day with SI. Even though this is a medical emergency, there are no fast-acting treatments available.

Ketamine is a medication that is commonly used to safely sedate children who require painful procedures in the emergency department. For nearly ten years, intravenous ketamine has also been shown to rapidly reduce SI in adults. However, ketamine as a treatment for SI has never been studied in adolescents. The primary study objective is to pilot a clinical trial that investigates intravenous ketamine to emergently treat SI in adolescents.

If intravenous ketamine can relieve symptoms of SI for youth, this would have tremendous effects on patients and would dramatically change how physicians treat adolescent mental health emergencies. If ketamine is effective for several weeks, as it is in adults, it will help temporize patients until they receive more long-term psychiatric care. At the system level, it has the potential to reduce emergency visits and lengthy admissions. The investigators feel that the results of this study will be generalizable to pediatric centres across Canada and beyond.

DETAILED DESCRIPTION:
Suicidal ideation (SI) is a common and often severe cause of morbidity in adolescents. Patients frequently present to the emergency department (ED) with severe and distressing thoughts of self-harm or suicide, and yet, there is currently no acute therapeutic intervention to offer them. The standard of care for patients who do not require admission is to discharge them home with resources for websites, apps, or telephone help lines. These interactions fail to address the underlying suicidal thoughts and leave patients, families and providers feeling very dissatisfied. Medications are nearly never initiated in the ED and patients who are already taking anti-depressants experience a very slow therapeutic onset, and often with unfavourable side effects that make medication compliance difficult and sometimes impossible.

For nearly ten years, intravenous ketamine has been shown to be an efficacious acute therapy in adult patients with suicidal ideation. A single dose of intravenous (IV) ketamine can rapidly reduce the severity of suicidal ideation by moderate to large effect sizes (Cohen's d = 0.5-0.8) during an ED visit, in an adult population. However, it has never been studied in a pediatric population. The study primary objective is to determine the feasibility of conducting a trial that investigates the efficacy of IV ketamine to reduce suicidal ideation in adolescents in the pediatric emergency department.

If intravenous ketamine can rapidly alleviate the severity of SI for adolescents, this would have tremendous effects on patients and families and dramatically change how ED physicians treat pediatric mental health emergencies. It would increase patient safety, reduce patient distress, morbidity, possibly mortality and alleviate family stress. If the therapeutic effect of ketamine is maintained for several days, as it is in adults, it will help temporize patient symptoms while they are connected with more long-term psychiatric care. At the system level, it may reduce rates of ED visits and, often lengthy, admissions to hospital. The investigators feel that the results of this study will be generalizable to pediatric centres across Ontario, Canada and beyond.

ELIGIBILITY:
Inclusion Criteria

1. Responds "yes" to ASQ questionnaire at triage, which asks; "Are you having thoughts of killing yourself right now?"
2. Moderate to severe suicidal ideation, defined as score ≥ 3 on the first 5 questions of the Beck Scale for Suicidal Ideation (SSI5)
3. Age 12 to 17 years, inclusive
4. Medically clear, as judged by the treating physician
5. Speaks English or French

Exclusion Criteria

1. Acute intoxication
2. Previously enrolled in the current study or another clinical trial
3. History of intellectual disability or autism spectrum disorder by patient/parent report
4. Active, or history of, psychosis or psychotic disorder
5. History of non-psychiatric neurologic disorder (e.g., epilepsy)
6. Any of the following contraindications to ketamine based on the drug monograph:

   1. Known allergy or hypersensitivity to ketamine by patient history
   2. History of cerebrovascular accident (stroke or aneurysm)
   3. History of elevated intracranial pressure or idiopathic intracranial hypertension
   4. Significant hypertension requiring daily medication
   5. Severe cardiac decompensation
7. On a Form 1
8. Requires physical or chemical restraint
9. History of violence while in hospital
10. Assessment by a mental health practitioner during the current ED visit prior to study enrollment
11. Pregnant or breastfeeding

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the study as measured by the percentage of eligible of patients able to complete the study protocol. | Baseline
  Data analysis for feasibility will be descriptive in nature and there will be no formal hypothesis testing. The percentage of eligible patients who complete the study will be reported.

SECONDARY OUTCOMES:
Baseline distribution of responses to the first 5 questions of Beck Scale for Suicidal Ideation (SSI5) | Baseline
  Estimates of central tendency (mean) and variance (standard deviation) from participant responses to the SSI5 at baseline will be measured and reported. These parameters will aid with sample size estimates for the larger definitive trial.
  The first 5 questions of Beck Scale for Suicidal Ideation (SSI5) is a five item questionnaire scored from 0 to 10, with higher scores indicating more severe suicidal ideation.
Baseline distribution of responses to the suicide item (#10) from the Montgomery-Asberg Depression Rating Scale (MARDS10) | Baseline
  Estimates of central tendency (mean) and variance (standard deviation) from participant responses to the MADRS10 at baseline will be measured and reported. These parameters will aid with sample size estimates for the larger definitive trial.
  The MADRS is a 10 item, 6-point, depression scale. Item 10 rates suicidal ideation from 0 (Enjoys life or takes it as it comes), to 6 (Explicit plans for suicide when there is an opportunity. Active preparations for suicide) with higher scores indicating more severe suicidal ideation.
Baseline distribution of responses to the suicide item (#9) from the Beck Depression Index (BDI9). | Baseline
  Estimates of central tendency (mean) and variance (standard deviation) from participant responses to the BDI9 at baseline will be measured and reported. These parameters will aid with sample size estimates for the larger definitive trial.
  The Beck Depression Inventory is a 21 item depression questionnaire. Item 9 rates suicidal ideation from 0 (I don't have thoughts of killing myself) to 3 (I would kill myself if I had the chance) with higher scores indicating more severe suicidal ideation.
Baseline pragmatic assessment of the first 5 questions of the Beck Scale for Suicidal Ideation (SSI5), the suicide item (#10) from the Montgomery-Asberg Depression Rating Scale (MADRS10), and the suicide item (#9) from the Beck Depression Index (BDI9). | Baseline
  Pragmatic assessment of the tool validity by asking each participant, which of the three tools best captures how they are feeling at baseline.
Blinding assessment | Baseline
  Blinding adequacy will be measured by asking each participant which intervention they think they received at the end of the 40 minute study drug infusion.
Treatment efficacy measured by the Beck Scale for Suicidal Ideation (SSI5) | 40 minutes post treatment start
  Suicidal ideation severity at the end of the 40-minute medication infusion will be measured using SSI5.
  The first 5 questions of Beck Scale for Suicidal Ideation (SSI5) is a five item questionnaire scored from 0 to 10, with higher scores indicating more severe suicidal ideation.
Treatment efficacy measured by the suicide item (#10) from the Montgomery-Asberg Depression Rating Scale (MARDS10) | 40 minutes post treatment start
  Suicidal ideation severity at the end of the 40-minute medication infusion will be measured using MADRS10.
  The MADRS is a 10 item, 6-point, depression scale. Item 10 rates suicidal ideation from 0 (Enjoys life or takes it as it comes), to 6 (Explicit plans for suicide when there is an opportunity. Active preparations for suicide) with higher scores indicating more severe suicidal ideation.
Treatment efficacy measured by the suicide item (#9) from the Beck Depression Index (BDI9) | 40 minutes post treatment start
  Suicidal ideation severity at the end of the 40-minute medication infusion will be measured using BDI9.
  The Beck Depression Inventory is a 21 item depression questionnaire. Item 9 rates suicidal ideation from 0 (I don't have thoughts of killing myself) to 3 (I would kill myself if I had the chance) with higher scores indicating more severe suicidal ideation.
Treatment durability measured by the Beck Scale for Suicidal Ideation (SSI5) | 80 minutes, 120 minutes, 24 hours, and seven days post treatment start
  The durability of a treatment effect on suicidal ideation will be measured by SSI5 at 80 minutes, 120 minutes, 24 hours, and seven days post treatment start.
  The first 5 questions of Beck Scale for Suicidal Ideation (SSI5) is a five item questionnaire scored from 0 to 10, with higher scores indicating more severe suicidal ideation.
Treatment durability measured by the suicide item (#10) from the Montgomery-Asberg Depression Rating Scale (MARDS10) | 80 minutes, 120 minutes, 24 hours, and seven days post treatment start
  The durability of a treatment effect on suicidal ideation will be measured by MADRS10 at 80 minutes, 120 minutes, 24 hours, and seven days post treatment start.
  The MADRS is a 10 item, 6-point, depression scale. Item 10 rates suicidal ideation from 0 (Enjoys life or takes it as it comes), to 6 (Explicit plans for suicide when there is an opportunity. Active preparations for suicide) with higher scores indicating more severe suicidal ideation.
Treatment efficacy measured by the suicide item (#9) from the Beck Depression Index (BDI9) | 80 minutes, 120 minutes, 24 hours, and seven days post treatment start
  The durability of a treatment effect on suicidal ideation will be measured by BDI9 at 80 minutes, 120 minutes, 24 hours, and seven days post treatment start.
  The Beck Depression Inventory is a 21 item depression questionnaire. Item 9 rates suicidal ideation from 0 (I don't have thoughts of killing myself) to 3 (I would kill myself if I had the chance) with higher scores indicating more severe suicidal ideation.
Admission to Hospital | 18 months
  The number and percentage of patients who require hospital admission at the enrolment ED visit will be reported.
Length of Stay in Hospital | 18 months
  The mean and standard deviation of length of hospital stay for patients admitted at the enrolment visit will be reported.
Revisits to the ED | 18 months
  The number and percentage of patients who require a repeat ED visit(s) for mental health complaints within 30 days following enrolment will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- CHEO, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schlegelmilch M, Plint AC, Barrowman N, Gray C, Bhatt M. Intravenous ketamine for emergency department treatment of suicidal ideation in a paediatric population: protocol for a double-blind, randomised, placebo-controlled, parallel-arm pilot trial (KSI study). BMJ Open. 2024 Jul 5;14(7):e085681. doi: 10.1136/bmjopen-2024-085681. PMID 38969374